CLINICAL TRIAL: NCT00937742
Title: The Effect of Processed Tomatoes on Endothelium- and Platelet- Function
Brief Title: The Effect of Processed Tomato Products on CVD Risks
Acronym: TOMATO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Tomato Products Wellness Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKE TOMATO
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Cardiovascular Disease
Keywords: cardiovascular disease; Lycopene; Tomato
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Non-tomato products (Experimental): Non-tomato products (i.e. teriyaki marinade, sprite, applesauce) to be consumed daily in replace of tomato products
  Interventions: Dietary Supplement: Tomato products

INTERVENTIONS:
Dietary Supplement: Tomato products — Specified amounts of tomato products (i.e. tomato juice, ketchup, salsa, tomato soup, spaghetti sauce) to be consumed daily during a 6 week intervention phase.

SUMMARY:
The primary working hypothesis is that consuming processed tomatoes frequently/daily will favorably improve endothelium and platelet function disease-risk biomarker profiles in adult men and women compared to consuming no or relatively low amounts of processed tomatoes.

ELIGIBILITY:
Inclusion Criteria:

men and women (>21 <70 years) nonsmokers, with a body mass index (BMI) ranging of 25 to 35 kg/m2, BP < or = 140/90 mmHg

Exclusion Criteria:

1. Total cholesterol (TC) is greater than 300 mg/dL;
2. Fasting triglyceride is greater than 300 mg/dL;
3. LDL cholesterol (LDL-C) is greater than 180 mg/dL;
4. Female subjects who are pregnant or lactating;
5. Subjects who are actively losing weight or trying to lose weight;
6. Subjects with known allergy or intolerance to tomato products;
7. taking any medications that would interfere with outcomes of the study, ie. lipid lowering medications, anti-inflammatory drugs, dietary supplements, such as fish oil or evening primrose;
8. subjects' with documented atherosclerotic disease, inflammatory disease, diabetes mellitus, uncontrolled hypertension (>=140/90 mm Hg - ok if controlled below this limit with medication), or other systemic diseases;
9. subjects with low hematological counts as determined by >or <15% the upper or lower cut-off values of normal established for the lab;
10. Smokers. -

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-01; Primary Completion 2008-09 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Platelet and monocyte function/activity | Baseline and end of intervention phase (week 6)
Vascular function | Baseline and end of intervention phase (week 6)

SECONDARY OUTCOMES:
Lipids | Baseline and end of intervention phase (week 6)
Insulin/Glucose | Baseline and end of intervention phase (week 6)
Inflammatory Markers | Baseline and end of intervention phase (week 6)

CONTACTS AND LOCATIONS:
Overall Officials: Penny M Kris-Etherton, PhD, Principal Investigator — Penn State University
Locations (1):
- Penn State University, University Park, Pennsylvania, United States